CLINICAL TRIAL: NCT04541043
Title: An Open-Label Extension (OLE) Study to Evaluate the Efficacy and Safety of Nefecon Treatment in Patients With IgA Nephropathy Who Have Completed Study Nef-301
Brief Title: Efficacy and Safety in Patients With Primary IgA Nephropathy Who Have Completed Study Nef-301 (Nefigard-OLE)
Acronym: Nefigard-OLE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Calliditas Therapeutics AB (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Nef-301 OLE; 2020-003308-14 (EudraCT Number)
Record Dates: First submitted 2020-09-01; First posted 2020-09-09 (Actual); Results first posted 2025-01-03 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2024-12

CONDITIONS: Primary IgA Nephropathy
MeSH Terms: conditions — Glomerulonephritis, IGA

STUDY DESIGN:
Intervention Model Description: This is an open label, single-arm study with active treatment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Active Nefecon treatment (Experimental): Nefecon 16 mg once daily by mouth for 9 months
  Interventions: Drug: Nefecon 16mg daily

INTERVENTIONS:
Drug: Nefecon 16mg daily — All study patients received Nefecon 16 mg daily for 9 months.

SUMMARY:
This is a Phase 3b, multicenter, open-label extension (OLE) study to evaluate the efficacy and safety of Nefecon treatment in patients with IgAN who have completed the Phase 3 Study Nef-301 and continue to be treated with a stable dose of RAS inhibitor therapy (ACEIs and/or ARBs). Patients who previously received Nefecon in Study Nef-301 will receive retreatment, whereas patients who previously received placebo in Study Nef-301 will be treatment naïve to Nefecon.

DETAILED DESCRIPTION:
This is a Phase 3b, multicenter, open-label extension (OLE) study to evaluate the efficacy and safety of Nefecon treatment in patients with IgAN who have completed the Phase 3 Study Nef 301 and continue to be treated with a stable dose of RAS inhibitor therapy (ACEIs and/or ARBs). Patients who previously received Nefecon in Study Nef-301 will receive retreatment, whereas patients who previously received placebo in Study Nef-301 will be treatment naïve to Nefecon. During Study Nef-301 OLE, the patients and Investigators will remain blinded to treatment given in Study Nef-301.

During Study Nef-301 OLE, patients will receive Nefecon for a 9-month period. The dose may be reduced if clinically relevant adverse events (AEs) develop during the 9-month Treatment Period that the Investigator considers related to the study drug and that mandate dose reduction.

Patients will remain on a stable dose of RAS inhibitor therapy (ACEIs and/or ARBs) throughout the study. The patient will come for a follow-up visit at 12 months after first dose.

ELIGIBILITY:
Inclusion Criteria:

1. Patients that completed study Nef-301
2. On a stable dose of RAS inhibitor therapy (ACEIs and/or ARBs) at the maximum allowed dose or maximum tolerated dose according to the 2012 KDIGO guidelines
3. Willing and able to provide written informed consent.
4. UPCR equal to or more than 0.8 g/gram
5. eGFR equal to or more than 30 mL/min per 1.73 m2 using the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) formula.

Exclusion Criteria:

1. Systemic diseases that may cause mesangial IgA deposition.
2. Patients who have undergone a kidney transplant;
3. Patients with presence of other glomerulopathies and/or nephrotic syndrome
4. Patients with acute, chronic, or latent infectious disease including hepatitis, tuberculosis (TB), human immunodeficiency virus (HIV), and chronic urinary tract infections;
5. Patients with liver cirrhosis, as assessed by the Investigator;
6. Patients with a diagnosis of type 1 or type 2 diabetes mellitus which is poorly controlled
7. Patients with history of unstable angina, class III or IV congestive heart failure, and/or clinically significant arrhythmia, as judged by the Investigator;
8. Patients with unacceptable blood pressure control defined as a blood pressure consistently above national guidelines for proteinuric renal disease, as assessed by the Investigator.
9. Patients with diagnosed malignancy within the past 5 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2020-11-17 (Actual); Primary Completion 2024-02-26 (Actual); Study Completion 2024-02-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Philipson, MD, Study Director — Calliditas Therapeutics AB
Locations (18):
- 13 Investigator sites, Palo Alto, California, United States
- 4 Investigator sites, Buenos Aires, Argentina
- 6 Investigator sites, Melbourne, Australia
- 3 Investigator sites, Minsk, Belarus
- 4 Investigator sites, Brussels, Belgium
- 7 Investigator sites, Québec, Canada
- 6 Investigator sites, Prague, Czechia
- 2 Investigator sites, Jyväskylä, Finland
- 2 Investigator sites, Saint-Priest-en-Jarez, France
- 5 Investigator sites, Aachen, Germany
- 5 Investigator sites, Athens, Greece
- 2 Investigator sites, Milan, Italy
- 2 Investigator sites, Lodz, Poland
- 4 Investigator sites, Gyeonggi-do, South Korea
- 4 Investigator sites, Barcelona, Spain
- 3 Investigator sites, Uppsala, Sweden
- 3 Investigator sites, Kayseri, Turkey (Türkiye)
- 6 Investigator sites, Leicester, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Retreatment - Previously Treated With Nefecon in Nef-301 Study; Delayed Treatment - Previously Treated With Placebo in Nef-301 Study: Nef-301-OLE study is an extension study to the Nef-301 study. Study results are analyzed based on treatment in the previous Nef-301 study where patients were randomized to receive either Nefecon or Placebo. Thus, in this Nef-301-OLE study the patients are either retreated with Nefecon or receiving Nefecon for the first time.
Period: Overall Study
Arm/Group | Retreatment - Previously Treated With Nefecon in Nef-301 Study | Delayed Treatment - Previously Treated With Placebo in Nef-301 Study
Started | 45 | 74
Completed | 43 | 62
Not Completed | 2 | 12

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Retreatment - Previously Treated With Nefecon in Nef-301 Study | Delayed Treatment - Previously Treated With Placebo in Nef-301 Study | Total
Number analyzed (Participants) | 45 | 74 | 119
Age, Continuous [Median (Full Range); unit: years] | 46 [29 to 70] | 47 [25 to 76] | 47 [25 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 19 | 25
  Male | 39 | 55 | 94
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 9 | 7 | 16
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 36 | 64 | 100
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 3 | 3
Region of Enrollment [Number; unit: participants]
  Argentina | 6 | 3 | 9
  Czechia | 2 | 13 | 15
  United States | 6 | 5 | 11
  United Kingdom | 3 | 3 | 6
  Belarus | 1 | 1 | 2
  Spain | 1 | 1 | 2
  Greece | 3 | 5 | 8
  Canada | 7 | 7 | 14
  South Korea | 2 | 4 | 6
  Sweden | 1 | 2 | 3
  Turkey | 0 | 2 | 2
  Belgium | 4 | 3 | 7
  Finland | 1 | 3 | 4
  Poland | 0 | 3 | 3
  Italy | 2 | 1 | 3
  Australia | 2 | 7 | 9
  France | 1 | 3 | 4
  Germany | 3 | 8 | 11
Urine Protein to Creatine Ratio (UPCR) [Geometric Mean (Inter-Quartile Range); unit: g/gram] | 1.253 [0.859 to 1.796] | 1.339 [1.000 to 1.881] | 1.306 [0.935 to 1.881]
Baseline Estimated glomerular filtration rate (eGFR) [Geometric Mean (Inter-Quartile Range); unit: ml/min/1.73 m2] | 51.0 [42.0 to 62.0] | 49.9 [39.9 to 64.9] | 50.3 [39.9 to 63.5]

OUTCOME MEASURES:

1. Primary Outcome: Ratio of Urine Protein to Creatine Ratio (UPCR) at 9 Months Compared to Baseline
Description: The outcome is measured as UPCR based on 24 hour urine collections at 9 months following the first dose of Nefecon compared to baseline Ratio being: UPCR at 9 months in g/gram divided with UPCR at Baseline in g/gram
Time Frame: 9 months
Population: Number of participants analyzed reflects number of patients with available data at baseline and 9 months .
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: ratio
Arm/Group | Retreatment - Previously Treated With Nefecon in Nef-301 Study | Delayed Treatment - Previously Treated With Placebo in Nef-301 Study
Number analyzed (Participants) | 44 | 69
ratio | 0.67 [0.56 to 0.80] | 0.69 [0.60 to 0.80]

2. Primary Outcome: Ratio of Estimated Glomerular Filtration Rate (eGFR) at 9 Months Compared to Baseline
Description: The outcome is measured as ratio of eGFR in mL/min/1.73 m2 (calculated using the CKD-EPI formula) at 9 months following the first dose of Nefecon compared to baseline. I.e. eGFR at 9 months divided by eGFR at Baseline.
Time Frame: 9 months
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: ratio
Arm/Group | Retreatment - Previously Treated With Nefecon in Nef-301 Study | Delayed Treatment - Previously Treated With Placebo in Nef-301 Study
Number analyzed (Participants) | 44 | 69
ratio | 0.97 [0.94 to 1.01] | 0.97 [0.94 to 1.00]

3. Secondary Outcome: Ratio of Urine Albumin to Creatinine Ratio (UACR) at 9 Months Compared to Baseline
Description: Ratio of urine albumin to creatinine ratio (UACR) measured by 24h urine sampling at 9 months compared to baseline. I.e. UACR at 9 months divided by eGFR at Baseline.
Time Frame: 9 months
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: ratio
Arm/Group | Retreatment - Previously Treated With Nefecon in Nef-301 Study | Delayed Treatment - Previously Treated With Placebo in Nef-301 Study
Number analyzed (Participants) | 44 | 69
ratio | 0.60 [0.49 to 0.75] | 0.65 [0.55 to 0.77]

4. Secondary Outcome: Change From Baseline Short Form 36 (SF-36) Quality of Life Assessment at 12 Months
Description: Short Form 36 (SF-36) quality of life assessment at 12 months compared to baseline, i.e. change from baseline.
  The 36-Item Short Form Health Survey (SF-36) is a set of generic, coherent, and easily administered quality-of-life measures. These measures rely upon patient self-reporting and have been widely used. It consists of eight health concepts: physical functioning, bodily pain, role limitations due to physical health problems, role limitations due to personal or emotional problems, emotional well-being, social functioning, energy/fatigue, and general health perceptions.
  Higher scores indicate better health. Scores represent the percentage of total possible score achieved, i.e. 0 is the minimum and 100 is the maximum score.
Time Frame: Baseline & 12 months
Measure: Mean (Standard Deviation); unit: Change in percentage of total Score
Arm/Group | Retreatment - Previously Treated With Nefecon in Nef-301 Study | Delayed Treatment - Previously Treated With Placebo in Nef-301 Study
Number analyzed (Participants) | 44 | 70
Change in percentage of total Score
  Bodily Pain | -4.518 (10.0522) | -3.756 (9.9213)
  General Health | -4.290 (7.4076) | -3.301 (5.8211)
  Mental Component Summary | -2.282 (7.1270) | -1.061 (6.6251)
  Mental Health | -1.725 (7.1576) | -1.570 (6.3522)
  Physical Component Summary | -3.952 (6.6367) | -3.403 (6.1115)
  Physical Functioning | -2.697 (7.4670) | -1.996 (6.6726)
  Role Emotional | -2.928 (7.2390) | -0.747 (7.4962)
  Role Physical | -3.421 (7.1914) | -2.793 (7.6901)
  Social Function | -4.102 (8.4631) | -2.364 (6.3713)
  Vitality | -2.633 (7.6406) | -2.376 (7.6968)

5. Secondary Outcome: Number of Patients With Microhematuria at 9 Months Compared to Baseline
Time Frame: 9 months
Measure: Count of Participants; unit: Participants
Arm/Group | Retreatment - Previously Treated With Nefecon in Nef-301 Study | Delayed Treatment - Previously Treated With Placebo in Nef-301 Study
Number analyzed (Participants) | 44 | 68
Participants | 10 | 17

6. Secondary Outcome: Number of Patients Receiving Rescue Treatment
Description: Systemic immunosuppressive drugs (including glucocorticoids in some situations ), dialysis, and renal transplantation are considered as rescue medications in this study.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Retreatment - Previously Treated With Nefecon in Nef-301 Study | Delayed Treatment - Previously Treated With Placebo in Nef-301 Study
Number analyzed (Participants) | 45 | 74
Participants | 1 | 0

7. Secondary Outcome: Proportion of Patients on Dialysis, Undergoing Kidney Transplantation, or With eGFR <15 mL/Min Per 1.73 m2
Description: Looking at number of patients with end stage kidney disease defined as being on dialysis, undergoing kidney transplantation, or having eGFR <15 mL/min per 1.73 m2
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Retreatment - Previously Treated With Nefecon in Nef-301 Study | Delayed Treatment - Previously Treated With Placebo in Nef-301 Study
Number analyzed (Participants) | 45 | 74
Participants | 2 | 0

8. Secondary Outcome: Change From Baseline Cortisol Suppression at 9 Months
Description: Cortisol suppression at 9 and 12 months, measured as urinary cortisol excretion over 24 hours compared to baseline.
Time Frame: Baseline & 9 months
Measure: Mean (Standard Deviation); unit: ug/day)
Arm/Group | Retreatment - Previously Treated With Nefecon in Nef-301 Study | Delayed Treatment - Previously Treated With Placebo in Nef-301 Study
Number analyzed (Participants) | 44 | 66
ug/day) | -24.122 (25.1690) | -32.126 (30.6978)

9. Secondary Outcome: Change From Baseline Cortisol Suppression at 12 Months
Description: Cortisol suppression at 9 and 12 months, measured as urinary cortisol excretion over 24 hours compared to baseline.
Time Frame: Baseline & 12 months
Measure: Mean (Standard Deviation); unit: ug/day
Arm/Group | Retreatment - Previously Treated With Nefecon in Nef-301 Study | Delayed Treatment - Previously Treated With Placebo in Nef-301 Study
Number analyzed (Participants) | 41 | 63
ug/day | -7.660 (27.4262) | -11.954 (25.8052)

ADVERSE EVENTS:
Time Frame: All-Cause Mortality, SAEs and non-serious AEs were assessed from date of first dose of study treatment until 12 months after the first dose of study drug.
Description: All-Cause Mortality, SAEs and non-serious AEs were assessed from date of first dose of study treatment until 12 months after the first dose of study drug.
Arm/Group | Retreatment - Previously Treated With Nefecon in Nef-301 Study | Delayed Treatment - Previously Treated With Placebo in Nef-301 Study
All-Cause Mortality (participants affected / at risk) | 0/45 | 0/74
Serious Adverse Events (participants affected / at risk) | 5/45 | 5/74
Other Adverse Events (participants affected / at risk) | 32/45 | 46/74
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Retreatment - Previously Treated With Nefecon in Nef-301 Study (N=45) | Delayed Treatment - Previously Treated With Placebo in Nef-301 Study (N=74)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Monoclonal B-cell lymphocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Joint dislocation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Scapula fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Central nervous system vasculitis (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Chorioretinopathy (Eye disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Retreatment - Previously Treated With Nefecon in Nef-301 Study (N=45) | Delayed Treatment - Previously Treated With Placebo in Nef-301 Study (N=74)
Corona virus infection (Infections and infestations) | 12 (12) | 13 (14)
Folliculitis (Infections and infestations) | 0 (0) | 4 (4)
Nasopharyngitis (Infections and infestations) | 1 (1) | 4 (4)
Upper respiratory tract infection (Infections and infestations) | 3 (3) | 2 (3)
Nausea (Gastrointestinal disorders) | 3 (3) | 2 (3)
Hypertension (Vascular disorders) | 8 (9) | 12 (13)
Acne (Skin and subcutaneous tissue disorders) | 3 (4) | 6 (7)
Weight increased (Investigations) | 3 (3) | 8 (8)
Fatigue (General disorders) | 4 (4) | 2 (2)
Oedema peripheral (General disorders) | 1 (1) | 10 (12)
Pyrexia (General disorders) | 0 (0) | 4 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (4) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 3 (4)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 6 (8) | 5 (6)
Insomnia (Psychiatric disorders) | 3 (3) | 6 (6)
Headache (Nervous system disorders) | 4 (6) | 3 (3)
Proteinuria (Renal and urinary disorders) | 4 (4) | 5 (5)
Cushingoid (Endocrine disorders) | 2 (2) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-08-06): https://cdn.clinicaltrials.gov/large-docs/43/NCT04541043/Prot_SAP_000.pdf